CLINICAL TRIAL: NCT06041035
Title: A Phase IB/II Clinical Study to Assess the Efficacy and Safety of QLS31905 in Combination With Chemotherapy as First-line Treatment in Patients With Claudin 18.2 (CLDN18.2) Positive Advanced Malignant Solid Tumors
Brief Title: A Study of QLS31905 Combination Chemotherapy as First-Line Treatment in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QLS31905-201
Record Dates: First submitted 2023-08-30; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Solid Tumor
Keywords: CLDN18.2; QLS31905
MeSH Terms: interventions — Taxes; Gemcitabine; Oxaliplatin; Capecitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- QLS31905 + nab-paclitaxel + gemcitabine (Part A/B) (Experimental): Pancreatic cancer participants will be treated with QLS31905 in combination with nab-paclitaxel and gemcitabine for part A of the study to establish the recommended dose of QLS31905 for part B. In part B, the participants will be treated with QLS31905 at a dose determined by the part A of the study in combination with nab-paclitaxel and gemcitabine.
  Interventions: Drug: QLS31905; Drug: Nab paclitaxel; Drug: Gemcitabine
- QLS31905 + oxaliplatin + capecitabine (Part B) (Experimental): In part B, gastric/gastroesophageal junction cancer participants will be treated with QLS31905 at dose determined by part A of the study in combination with oxaliplatin and capecitabine.
  Interventions: Drug: QLS31905; Drug: Oxaliplatin; Drug: Capecitabine
- QLS31905 + gemcitabine+cisplatin(Part B) (Experimental): In part B, other solid tumor participants including but not limited to biliary tract cancer will be treated with QLS31905 at dose determined by part A in combination with standard chemotherapy recommended by guidelines.QLS31905 plus gemcitabine+ cisplatin as the first-line treatment of advanced biliary tract cancer.
  Interventions: Drug: QLS31905; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: QLS31905 — Administered as an intravenous infusion.
Drug: Nab paclitaxel — 125 mg/m2 administered as IV infusion on D1/D8/D15 of each cycle.
  Arms: QLS31905 + nab-paclitaxel + gemcitabine (Part A/B)
Drug: Gemcitabine — 1000 mg/m2 administered as IV infusion on D1/D8/D15 of each cycle.
  Arms: QLS31905 + gemcitabine+cisplatin(Part B); QLS31905 + nab-paclitaxel + gemcitabine (Part A/B)
Drug: Oxaliplatin — 85 mg/m2, intravenous infusion, D1/D15, up to 6 cycles.
  Arms: QLS31905 + oxaliplatin + capecitabine (Part B)
Drug: Capecitabine — 1000 mg/m2, oral, bid, D1-D7,D15-D21, up to 6 cycles.
  Arms: QLS31905 + oxaliplatin + capecitabine (Part B)
Drug: Cisplatin — 25 mg/m2, intravenous infusion, D1/D15, up to 6 cycles.
  Arms: QLS31905 + gemcitabine+cisplatin(Part B)

SUMMARY:
This study aims to evaluate the efficacy and safety of QLS31905 plus chemotherapy in patients with Claudin18.2-positive advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in the study and sign the informed consent form;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1;
* Expected survival time ≥ 3 months;
* Histologically or cytologically confirmed locally advanced unresectable or metastatic solid tumors;
* No prior systemic anti-tumor treatment for locally advanced unresectable or metastatic disease;
* Tumor tissue samples determined to have moderate-to-high Claudin18.2 expression by immunohistochemistry (IHC);
* At least one measurable lesion per RECIST v1.1;
* Patients with adequate cardiac, liver, renal function, etc.

Exclusion Criteria:

* History of malignancies other than the target cancer within 5 years prior to the first dose of the investigational product ;
* Underwent major organ surgery (excluding needle biopsy) or had significant trauma within 28 days prior to enrollment, or requires elective surgery during the study;
* Known central nervous system metastases;
* Patients with hepatitis B; patients with hepatitis C; patients who test positive for syphilis, or patients with a known history of HIV or positive HIV screening test;
* Patients with a known history of psychoactive drug abuse, alcohol abuse, or substance abuse;
* Patients with added risks associated with the study or may interfere with the interpretation of study results as determined by the investigator, or deemed unsuitable by the investigator and/or sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) (Part A) | Approximately 12 months
  As measured by number of participants experiencing dose related toxicity (DLT) in each escalating cohort.
Phase 2 Recommended Dose（RP2D)(Part A) | Approximately 12 months
  Monitor for MTD, and minimal efficacious dose by monitoring responses at different dose levels.
Objective response rate (ORR)(Part B) | Approximately 12 months
  ORR is defined as the proportion of participants who have a best overall response of Complete Response (CR) or Partial Response (PR) as assessed by investigator evaluation per RECIST 1.1.

SECONDARY OUTCOMES:
Safety assessed by Adverse Events (AEs) | Approximately 12 months
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom,or disease (new or exacerbated) temporally associated with the use of a medicinal product.
Safety assessed by incidence of serious adverse events (SAE) | Approximately 12 months
  Adverse Event (AE) is considered "serious" if the investigator or sponsor view any of the following outcomes: Death, life-threatening, persistent or significant disability/incapacity, congenital anomaly or birth defect,hospitalization, or medically important event.
Number of participants with laboratory value abnormalities and/or adverse events (AEs) | Approximately 12 months
  Number of participants with potentially clinically significant laboratory values.
Progression Free Survival(PFS) | Approximately 12 months
  PFS is defined as the duration from the subject's first dose of the investigational product to the first imaging confirmation of progressive disease per RECIST 1.1 by investigator evaluation or death due to any cause (whichever occurs first).
Duration Of Response (DOR) | Approximately 12 months
  DOR is defined as the time from the date of the first response (CR/PR) until the date of progressive disease as assessed by investigator evaluation per RECIST 1.1 or death due to any cause (whichever occurs first).
Overall Survival (OS) | Approximately 12 months
  OS is defined as the duration from the first dose of the investigational product to the time point when death occurs due to any cause.
Pharmacokinetics(PK) of QLS31905: Maximum concentration (Cmax) | Approximately 12 months
  Cmax will be derived from the PK serum samples collected.
PK of QLS31905: Time of the maximum concentration (Tmax) | Approximately 12 months
  Tmax will be derived from the PK serum samples collected.
PK of QLS31905: Terminal elimination half-life (T1/2) | Approximately 12 months
  T1/2 will be derived from the PK serum samples collected.
PK of QLS31905: Clearance (CL) | Approximately 12 months
  CL will be derived from the PK serum samples collected.
PK of QLS31905: Apparent volume of distribution during the terminal phase (Vz) | Approximately 12 months
  Vz will be derived from the PK serum samples collected.
Number of anti-drug antibody (ADA) Positive Participants | Approximately 12 months
  Immunogenicity will be measured by the number of participants that are ADA positive.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China